CLINICAL TRIAL: NCT06962111
Title: Early-Stage Partner in Care-Living Alone (EPIC-LA)
Brief Title: Early-Stage Partner in Care Living Alone Plus
Acronym: EPICLA+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Abigail Gomez Morales, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00020497; 1P30AG086561 (NIH)
Record Dates: First submitted 2025-03-31; First posted 2025-05-08 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-03

CONDITIONS: Dementia; Mild Cognitive Impairment (MCI); Alzheimer Disease
Keywords: Living Alone; Memory Disorders; Older adults (60 years and older); Alzheimer Disease and Related Dementias; Early Stage Alzheimer disease; Intervention; Skill-building
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Alzheimer Disease; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (assigned by chance) to one of two groups: 1) EPICLA+ or 2) Wait List Control (WLC).
  The WLC group is offered EPICLA+ after the T2. For the WLC, comparing their T2 and T3 assessments provides an opportunity to examine within-person change before and after receiving the EPICLA+ intervention. For those assignments at T1 to EPIC LA+, follow-ups between T2 and T3 provide opportunities to examine maintenance of gains.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EPICLA+ (Experimental): Group EPICLA+ will start the intervention immediately after assessment 1. The EPICLA+ program consists of a 7-session, psychoeducational skills training intervention, held via Zoom, designed to assist people with early-stage memory loss that live alone in the community by providing early-stage-related education and skill-training sessions to reduce stress, enhance well-being, manage challenges, and plan for the future. Following the 7 EPIC sessions, participants will attend a booster session, held via Zoom, to reinforce the skills/lessons.
  Interventions: Behavioral: Psychoeducational skills training intervention
- Wait List Control (WLC) (Active Comparator): The WLC group will start the intervention after 3 months of the EPICLA+ group start date, once T2 assessment is completed.
  Interventions: Behavioral: Psychoeducational skills training intervention

INTERVENTIONS:
Behavioral: Psychoeducational skills training intervention — This protocol is a minimal risk care values clarification /care planning and psychoeducational skills training intervention, delivered as a workshop series plus one in-home session for people in the early stages of memory loss who live alone. In addition, during this intervention, participants will have access to general and personalized virtual resources with materials for use during and after the intervention.

SUMMARY:
EPICLA+ (Early-Stage Partners in Care Living Alone Plus) is a research project designed to assist people with early-stage memory loss who live alone in the community by providing early-stage related education and skill-training sessions, held via Zoom, designed to reduce stress, enhance well-being, manage challenges, and plan for the future. Researchers will gather feedback from individuals about their experience to continue to improve programs for early-stage memory loss.

DETAILED DESCRIPTION:
This study aims to create a supportive environment to help individuals with early-stage memory loss or early-stage dementia living alone in the community by providing education and skill-training programs, held via Zoom, where they can be educated in memory changes associated with dementia, learn to manage behavioral changes, improve communication skills, cope with stress, and plan for the future. About 70 people will be enrolled across the United States through Arizona State University.

People who decide to participate in this program voluntarily will be asked to:

Meet others in the earlier stages of memory loss who live alone Attend six group sessions via Zoom (2 hours and 30 minutes each) to learn strategies for handling new situations, reducing stress, improving mood, communicating better with others, and planning for the future.

Participate in one 90-minute individualized session via Zoom to address specific issues unique to each one's situation.

Participate in three 45-minute confidential interviews that involve questions about background, mood, and quality of life.

Participate in a booster session for those initially assigned to EPICLA+, lasting approximately 2h 30 minutes.

Participate in interviews at the start, and again about 3 and 6 months, via Zoom, to help us continue to improve the program.

All participants are offered the EPICLA+ sessions shortly after their first interview or shortly after their 3-month interview.

ELIGIBILITY:
Early-stage inclusion criteria

1. Must be at least 60 years of age
2. Must be able to participate in English or Spanish
3. Must be a US resident
4. Must be able to provide consent verbally and in writing (electronically or via mail)
5. Must exhibit at least 2 of 8 changes caused by thinking and memory problems on the AD8 (a reliable and valid 8-item dementia screening tool).
6. The Early-stage individual must have a diagnosis of early-stage ADRD or have a Mini-Mental State Exam (MMSE) score:

   1. between 20-26 for those who have completed high school, or
   2. between 17-26*, for those who have not completed high school, or
   3. 27 or higher with a confirmed diagnosis of early-stage dementia or MCI.
7. Able to participate in EPIC-LA workshops via zoom

   Exclusion Criteria:
8. Inability to participate via telephone or online video conferencing service.
9. The participant expresses feelings of not wanting to participate
10. The participant do not have enough time to attend the training,
11. The participant demonstrates lack of skills with using a computer that precludes participation
12. The participant does not have a stable internet connection to connect to the video platform
13. The participant has difficulty hearing or a visual impairment that precludes participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Quality of Life in Alzheimer's Disease (QoL-AD) | Baseline, at 3 months, and at 6 months
  This scale assesses 13 global items of quality of life covering areas like physical health, mood, family, and finances, with the outcomes poor, fair, good, and excellent. It can be used across different dementia stages and is designed for individuals with dementia and their caregivers. The scale consists of 13 questions. Each question has four possible responses - poor, fair, good, and excellent, each equating to 1-4 points respectively. The total score ranges from 13 to 52, with higher scores indicating a higher quality of life.
UCLA 3-item Loneliness Scale | Baseline, at 3 months, and at 6 months
  This scale comprises three questions that measure three dimensions of loneliness: relational connectedness, social connectedness, and self-perceived isolation. The scale is rated with hardly ever, some of the time, and often, with scores ranging from 1 to 3, respectively. The total score ranges from 3 to 9, with scores ranging from 6 to 9 indicating loneliness.
Dementia Quality of Life (DQoL)- Positive and Negative Feelings Affect Scale | Baseline, at 3 months, and at 6 months
  The DQoL consists of 30 items and five scales: positive affect (six items), negative affect (11 items), feelings of belonging (three items), self-esteem (four items), sense of aesthetics (five items) and one global item. QDOL is a Likert scale with the outcomes never, seldom, sometimes, often, and very often, ranging from 1 to 5, respectively. Higher scores indicate better QoL, except on the negative affect scale. The study focuses on assessing positive (e.g., content) and negative (e.g., afraid) feelings.
Center of Epidemiologic Studies-Depression short form (CES-D) | Baseline, at 3 months, and at 6 months
  Shortened version of the CESD-20. It measures depressive symptoms and assesses feelings such as feeling bothered by things, having trouble concentrating, etc. It is scored by summing the responses to its 10 items, each rated on a 4-point scale with scores rarely or none of the time, some of the time, occasionally, and most of the time, ranging from 0 to 3, respectively. Total scores range from 0 to 30, with higher scores indicating greater depressive symptoms.
Hopkins Symptoms Checklist - Anger Subscale | Baseline, at 3 months, and at 6 months
  Tool used for assessing feelings, such as feeling critical of others, irritated, tense, calm, etc., using the Likert scale not at all, a little, somewhat, and very much with scores ranging from 0 to 3 respectively. higher scores indicate higher levels of anger.

SECONDARY OUTCOMES:
Care Preparedness Scale | Baseline, at 3 months, and at 6 months
  Assessment of the level of preparedness associated with future care using the Likert scale: not at all prepared, not too well prepared, somewhat well prepared, pretty well prepared, and very well prepared. Scores range from 1 to 5. Higher scores indicate higher levels of care preparedness.
Leisure Satisfaction Scale | Baseline, at 3 months, and at 6 months
  Assessment of the diligence in one's own health and leisure activity satisfaction using the ratings not at all, a little, and a lot. Scores range from 1 to 3, respectively, with higher scores indicating higher levels of leisure satisfaction and diligence in one's own health.
Knowledge of Dementia (modified) | Baseline, at 3 months, and at 6 months
  Assessment of the knowledge and understanding of dementia, causes, course, and treatment. Answers are true or false.
Care preferences/circle diagrams | Baseline, at 3 months, and at 6 months
  Peferences for who (informal or paid help) assist with care. Choices are: care partner, family/friends and Paid helper.
Decision-making in daily and long-term care | Baseline, at 3 months, and at 6 months
  Discussion with others on daily and future care options. The answers to the choices are like it very much, like it somewhat, dislike it somewhat, dislike it very much, and don't know.
Emotional-Intimacy Disruptive Behavior Scale | Baseline, at 3 months, and at 6 months
  Assessment of the degree of communication and openness with others. Respondents rate the extent to which they engaged in the behavior using the ratings none of the time, some of the time, much of the time, and most or all of the time. Scores range from 1 to 5, respectively, with higher scores indicating higher engagement in disruptive behavior.
Dementia Quality of life Instrument- self-esteem subscale | Baseline, at 3 months, and at 6 months
  A subscale specifically designed to assess the level of confidence, accomplishment, and decision-making in people with dementia. The assessment is measured with the outcomes never, seldom, sometimes, often, and very often, with scores ranging from 1 to 5, respectively, with higher scores indicating higher levels of confidence.

OTHER OUTCOMES:
Mini-Mental State Examination (MMSE) | Baseline, at 3 months, and at 6 months
  Gives a brief assessment of mental state status. It assesses different aspects of cognitive function, including orientation, memory, language, and visuospatial skills through different activities. The test is scored out of 30, with lower scores indicating more significant cognitive impairment.
Socio-demographics | Screening and baseline
  Socio-demographics characteristics questions (e.g., level of education, marital status).
Perception of benefits and acceptability | At 3 months or at 6 months
  Perceived study benefits questions (e.g., How much do you think you benefitted from participating in EPIC Living Alone Plus?)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Gomez-Morales, Principal Investigator — ASU
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No